CLINICAL TRIAL: NCT01921842
Title: Promoting Nutrition and Physical Activity in Child Care Centers
Brief Title: Child Care Wellness Study on Nutrition and Physical Activity
Acronym: CCWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Yale University (Other); University of California, San Francisco (Other); HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-1861; R40MC08727 (Other Grant/Funding Number: Maternal and Child Health Bureau)
Record Dates: First submitted 2013-08-07; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition and Physical Activity Training (Experimental): NAP-SACC Child Care Wellness program administered in year 1 of study
  Interventions: Behavioral: NAP-SACC Child Care Wellness Program
- Delayed Intervention Group (Other): NAP-SACC Child Care Wellness Program is administered in year 2 of study.
  Interventions: Behavioral: NAP-SACC Child Care Wellness Program

INTERVENTIONS:
Behavioral: NAP-SACC Child Care Wellness Program — Nutrition And Physical activity Self-Assessment for Child Care

SUMMARY:
The study is an evaluation of a nutrition and physical activity intervention in child care centers in NC, CA, and CT.

DETAILED DESCRIPTION:
The broad, long term goal is to develop a reproducible nutrition and physical activity intervention which utilizes child care consultant nutrition specialists to reduce the risk of overweight among children in regulated out-of-home child care. The objectives are:

1. To train Child Care Health consultants (CCHCs) to become specialists in nutrition consultation in child care such that they will increase their daily consultation activities on nutrition, physical activity, and childhood overweight,
2. To increase child care staff and parental knowledge of and positive attitudes toward providing healthy foods, appropriate portions of foods, and appropriate levels of physical activity for young children in out-of-home child care centers.,
3. To strengthen child care center policies, procedures, practices and behaviors, regarding providing healthy foods, appropriate portions of foods, and appropriate levels of physical activity for young children in out-of-home child care centers, and
4. To improve dietary intake and levels of physical activity, and to prevent increases in overweight and the risk of overweight as determined by body mass indexes among children in out-of-home child care centers.

ELIGIBILITY:
Inclusion Criteria:

* In each of the three geographical areas (NC, CA, CT), two pairs of community-based child care centers in urban areas with English-speaking directors, kitchens, and with 50-60 children between the ages of 2 and 5 years, 35% of whom are eligible for subsidy.

Exclusion Criteria:

* If the randomly selected child care center has an open case of child abuse or neglect.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in Nutrition and Physical Activity Policies | Baseline, Year 1, Year 2
  Determine if the use of a Nurse Child Care Health Consultant changes nutrition and physical activity policies at child care centers using criteria based on the national standards identified from resources such as NAEYC accreditation guidelines, Child and Adult Care Food Program (CACFP) policies and requirements, and the joint APHA/AAP publication Caring for our Children (American Academy of Pediatrics, American Public Health Association & National Resource Center for Health and Safety in Child Care, 2002; 1992). If written policies were present, they were compared to the gold-standard criteria from the national resource material and assigned a rating of either none (no written policies), poor (written policies fail to meet either state regulatory criteria or national standards), adequate (meets state regulatory criteria but not all of the national standards), or excellent (meets all of the national criteria present).

SECONDARY OUTCOMES:
Change in Nutrition and Physical Activity Behaviors | Baseline, Year 1, Year 2
  Determine if the use of a Nurse Child Care Health Consultant changes nutrition and physical activity behaviors at child care centers using the NAP SACC instrument intervention tool which consists of fifteen different areas of interest (9 nutrition and 6 physical activity) with several items each. The total number of items scored, 34, evaluate the center's environment with regard to support of healthy eating and regular physical activity. The instrument scoring is at one of four levels moving from minimal to best practice.

OTHER OUTCOMES:
Change in Body-Mass Index (BMI) of children in child care centers | Baseline, Year 1, Year 2
  Determine if the use of a Nurse Child Care Health Consultant changes BMI of children at child care centers.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Kotch, MD, Principal Investigator — University of North Carolina in Chapel Hill
Locations (1):
- Child Care Centers, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Alkon A, Crowley AA, Neelon SE, Hill S, Pan Y, Nguyen V, Rose R, Savage E, Forestieri N, Shipman L, Kotch JB. Nutrition and physical activity randomized control trial in child care centers improves knowledge, policies, and children's body mass index. BMC Public Health. 2014 Mar 1;14:215. doi: 10.1186/1471-2458-14-215. PMID 24580983